CLINICAL TRIAL: NCT02116166
Title: Claude D. Pepper Older Americans Independence Center (OAIC); Skeletal Muscle Inflammation, Oxidative Stress and DNA Repair in Age-Related Sarcopenia
Brief Title: Skeletal Muscle Inflammation, Oxidative Stress and DNA Repair in Age-Related Sarcopenia
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 201300790-N; 2P30AG028740 (NIH)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Sarcopenia
Keywords: aging; sarcopenia; mitochondria; skeletal muscle; inflammation
MeSH Terms: conditions — Sarcopenia; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skeletal muscle biopsy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Young: Young (20-35 years old)
- Old: Older (70-99 years old)

SUMMARY:
The purpose of this research study is to investigate how and why the loss of muscle mass occurs with aging. Tissue collected from young subjects will be compared to previously collected tissue from elderly subjects, as well as previously collected data on muscle function/mass to further investigate cellular and molecular pathways that have recently been shown to be important for the aging process in muscle. The Principal Investigator (PI) and the study team will look for specific proteins (called biomarkers) that can be present in the muscle tissue in various amounts in different individuals. This study will increase the investigators understanding of the processes of muscle atrophy (loss of mass) and functional loss at older age and will help to find new treatments and interventions aimed at improving the quality of life and independence of America's rapidly expanding elderly population.

DETAILED DESCRIPTION:
For this project, we will continue to gain mechanistic insight into age-related muscle loss and to maximize the utility of the tissue we previously collected (Claude D. Pepper Older Americans Independence Center (OAIC); Skeletal muscle apoptosis and physical performance; Oxidative RNA/DNA damage and repair in aged human muscle (Developmental Study), IRB # 429-2005) and we will collect muscle tissue from additional young subjects. This project will specifically test whether inflammatory pathways and DNA repair mechanisms are altered and/or involved in the development of sarcopenia and the related decline in physical function observed in the elderly.

Aim 1. We will further determine the association of skeletal muscle mass and function with intramuscular mediators of inflammation. Focus will be on inflammatory proteins (e.g.,TNF, TNFR1, pIkBα, pIKKb, CCL2, ZIP14, ZnT2) and genes (e.g., IL-6, TNFa, IL11β, IL-8, CCL2, CCR2, NFkB p50, NFkB p65, ZIP14) and metals (e.g., copper, zinc, and iron). We hypothesize that the majority of these markers will be upregulated in muscle from older individuals when compared to young.

Aim 2. For the first time, we will determine the age related effect of DNA damage on pattern and dynamics of mRNA translation in human muscle tissue by genome wide analysis using "ribosome profiling." The recently developed deep-sequencing techniques of RNA-seq and "ribosome profiling" will be implemented on human muscle. This will allow us to explore on a genomic scale and at single-nucleotide resolution, the effect of age-related DNA damage on transcriptional fidelity and translational kinetics. Importantly, for the first time, these phenotype changes will be compared with genome mapping of DNA damage, a major factor driving mammalian aging. We hypothesize that older muscle has greater modification of translational patterns compared to young muscle.

Muscle tissue samples remaining following the completion of this research will be stored and used in the future to explore new avenues of research related to aging.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged 20-35.
* willing and able to give informed consent.

Exclusion Criteria:

* High physical activity level (i.e., the subject has spent greater than 300 minutes per week in the past 2 month performing structured physical activity, such as exercising at a gym and/or weight training)
* Active treatment for cancer or history of cancer in the past 3 years
* Congestive heart failure NYHA Class III or IV
* Previous stroke with upper and/or lower extremities involvement within the last 6 months
* Peripheral vascular disease Fontaine Class III/IV
* History of life-threatening cardiac arrhythmias, stroke, severe Parkinson's disease or severe neurological disorders likely to interfere with physical function
* Renal disease requiring dialysis
* Lung disease requiring steroids
* Lower extremity amputation
* Complicated diabetes
* Life-threatening illnesses with an estimated life expectancy less than 1 year
* Anticoagulant therapy (aspirin use is allowed, but participants will be asked to stop taking it 48 hours prior to muscle biopsy)
* Involved in active weight loss > 5 kg in prior 3 months
* Pregnancy (determined by a pregnancy test)
* Lidocaine allergy

Temporary exclusion criteria:

* Recent bacterial infection (< 2 weeks)
* Acute febrile illness in previous 2 months
* High blood pressure (i.e., BP ≥ 160/90 mm Hg) at the visit (subject will be referred to his/her physician and reevaluated after appropriated therapy being instituted)
* Taking aspirin within 48 hours preceding biopsy
* Performing exercise 48 hours prior to the biopsy.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young (age 20-35 years; N =10)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Tumor Necrosis Factor alpha (TNF-alpha) | baseline
  Inflammation marker; measured in muscle biopsy specimens.
tumor-necrosis factor receptor-1 (TNFR1) | baseline
  Inflammation marker; measured in muscle biopsy specimens.
Phospho-Inhibitory Subunit Of NF-KBα (pIkBα) | baseline
  Inflammation marker; measured in muscle biopsy specimens.
Chemokine (C-C motif) ligand 2 (CCL2) | baseline
  Inflammation marker; measured in muscle biopsy specimens.
zinc transporter (ZIP) 14 | baseline
  Inflammation marker; measured in muscle biopsy specimens.
Interleukin 6 (IL-6) | baseline
  Inflammation marker; measured in muscle biopsy specimens.
Interleukin (IL) 11β | baseline
  Inflammation marker; measured in muscle biopsy specimens.
Interleukin 8 (IL-8) | baseline
  Inflammation marker; measured in muscle biopsy specimens.
C-C chemokine receptor type 2 (CCR2) | baseline
  Inflammation marker; measured in muscle biopsy specimens.
zinc transporter 14 (ZIP14) | baseline
  Inflammation marker; measured in muscle biopsy specimens.
copper | baseline
  metals; measured in muscle biopsy specimens.
zinc | baseline
  metals; measured in muscle biopsy specimens.
iron | baseline
  metals; measured in muscle biopsy specimens.
ribosome profiling | baseline
  DNA damage on pattern and dynamics of mRNA translation in human muscle tissue; measured in muscle biopsy specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Leeuwenburgh, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- See also: University of Florida Claude D. Pepper Older Americans Independence Center (OAIC) — http://aging.ufl.edu/?q=pepper_center